CLINICAL TRIAL: NCT05737615
Title: A Phase I Study of Pretargeted PET Imaging Using 64Cu-Tz-SarAr and a Trans-Cyclooctene-Modified Humanized 5B1 Immunoconjugate (hu5B1-TCO) in Patients With Pancreatic, Bladder Cancer, Gastrointestinal Malignancies or Solid Tumors With Elevated CA19-9
Brief Title: PET Imaging Using 64Cu-Tz-SarAr and hu5B1-TCO in People With Pancreatic, Colorectal, Bladder Cancer or Cancers With Elevated CA19.9
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study tracer is currently unavailable
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20-409
Record Dates: First submitted 2023-02-10; First posted 2023-02-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Primary Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer
Keywords: Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Ductal Adenocarcinoma; Primary Pancreatic Ductal Adenocarcinoma; Metastatic Pancreatic Cancer; hu5B1-TCO; 64Cu-Tz-SarAr; 20-409; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Positron-Emission Tomography; Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Pancreatic Cancer (Experimental): Participants have histologically confirmed primary or metastatic pancreatic ductal adenocarcinoma
  Interventions: Diagnostic Test: PET Scan; Drug: hu5B1-TCO; Drug: 64Cu-Tz-SarAr; Diagnostic Test: Pharmacokinetics

INTERVENTIONS:
Diagnostic Test: PET Scan — Participants will be imaged up to 4 time points post-injection to allow for biodistribution and dosimetry determination
Drug: hu5B1-TCO — On study day 0, a single slow infusion of hu5B1-TCO will be administered intravenously. Subsequently, either 3 days (n = 3) or 5 days (n = 3) later, a single slow infusion of 64Cu-Tz-SarAr will be administered intravenously.
Drug: 64Cu-Tz-SarAr — On study day 0, a single slow infusion of hu5B1-TCO will be administered intravenously. Subsequently, either 3 days (n = 3) or 5 days (n = 3) later, a single slow infusion of 64Cu-Tz-SarAr will be administered intravenously.
Diagnostic Test: Pharmacokinetics — All participants receiving 64Cu-Tz-SarAr will have serial blood samples drawn.

SUMMARY:
The purpose of this study is to find the highest safe dose of hu5B1-TCO and the best dosing schedule of hu5B1-TCO and 64Cu-Tz-SarAr for finding cancer cells that are CA19-9 positive. This study will also help to find out how much radiation the body is exposed to when 64Cu-Tz-SarAr is used, and provide information on the way the body absorbs, distributes, and gets rid of 64Cu-Tz-SarAr.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible for enrollment if they fulfill the following criteria:

1. Signed informed consent
2. 18 years of age or older
3. Histologically confirmed primary or metastatic pancreatic ductal adenocarcinoma/bladder carcinoma / gastrointestinal tumor reviewed at MSK - includes patients with biopsy-proven or high suspicion on imaging for pancreatic ductal adenocarcinoma (PDAC) or histologically confirmed, locally-advanced, or metastatic pancreatic ductal adenocarcinoma (PDAC) of

Patient with solid tumors increased serum CA19-9 serum level greater than ULN or CA19-9 positive biopsy

4. At least one lesion by CT or MRI ≥ 2 cm unless determined otherwise for presurgery subjects 5. ECOG performance status of 0 to 2 6. Adequate laboratory parameters including: i. Absolute neutrophil count (ANC) ≥1.5 x 109/L ii. Hemoglobin ≥ 9.0 g/dL iii. Platelet count >75,000/ mm3 iv. AST/SGOT, ALT/SGPT ≤2.5 x ULN, unless liver metastases are clearly present, then ≤5.0 x ULN v. Total bilirubin ≤ 1.5x the upper limit of normal unless considered due to Gilbert's syndrome in which case, ≤3x the upper limit of normal vi. Creatinine clearance (CLcr) (> 60 mL/min) estimated by the Cockcroft-Gault (C-G) equation or estimated glomerular filtration rate (eGFR) 10. Willingness to participate in collection of pharmacokinetic samples

Exclusion Criteria:

Patients will be excluded from the study if they fulfill any of the following criteria:

1. Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
2. Major surgery other than diagnostic surgery within 4 weeks of Study Day 1
3. History of anaphylactic reaction to human, or humanized, antibody
4. Other on-going cancer therapy with investigational agents
5. Known history of HIV
6. Pregnant or currently breast-feeding

   a. Subjects and their partners with reproductive potential must agree to use an effective form of contraception during the study and for 1 week following the study treatment.
7. Psychiatric illness/social situations that would interfere with compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
SUV mean measurement | 28 months
  The serial quantitative data obtained over the various organs of interest (heart, liver, spleen, kidney, lung and any other organ that exhibits uptake) will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Somali Gavane, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org